CLINICAL TRIAL: NCT03112629
Title: IMPULSE Enhanced - Study to Improve Outcomes in Aortic Stenosis - International, Multi-centre, Prospective, Observational Cohort Study
Brief Title: Study to Improve Outcomes in Aortic Stenosis
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: Impulse enhanced
Record Dates: First submitted 2017-03-21; First posted 2017-04-13 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Aortic Valve Stenosis
Keywords: Quality of Care; aortic stenosis; transcatheter aortic valve implantation; surgical aortic valve replacement; facilitated data relay
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- symptomatic AS: Patients diagnosed with severe aortic stenosis in echocardiography who display one or more of the following symptoms: exertional shortness of breath, chest pain, exertional dizziness or syncope.
- asymptomatic AS: Patients diagnosed with severe aortic stenosis in echocardiography who do not display symptoms

SUMMARY:
Multi-centre, multi-national, observational, prospective registry in four central full access centres in Germany (2), France (1) and the United Kingdom (1) and up to two satellites per hub (smaller hospitals / office based cardiologists (OBC) without access to surgical and percutaneous aortic valve (AV) interventions).

The hypothesis is that the management of patients with severe AS will differ between sites with on-site access to all treatment modes and those without such facilities.

DETAILED DESCRIPTION:
Data from existing studies indicate that the treatment pathways for patients with severe aortic stenosis with or without symptoms are insufficiently defined. This lack of definition can contribute both to delay in treatment and inappropriate treatment decisions. While this has been confirmed in hospitals with a full complement of treatment modalities for severe aortic stenosis, including surgery and percutaneous options, it is not known whether delay in treatment or appropriateness of treatment decisions are better or worse in smaller hospitals without equivalent on-site access.

The aim of this study is to delineate the case load of patients with aortic stenosis, outline the management of these patients and determine appropriateness in participating centres with and without on-site access to surgery and percutaneous treatment.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* identified on echocardiography with severe aortic stenosis, defined as at least one of:
* aortic valve area < 1 cm2
* indexed valve area < 0.6 cm2/m2
* maximum jet velocity > 4.0 m/sec
* mean transvalvular gradient > 40 mmHg

Exclusion Criteria:

* non-severe aortic stenosis
* previous aortic valve repair

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults aged over 18years identified on echocardiography with severe AS (irrespective of symptoms).
Sampling Method: Non-Probability Sample
Enrollment: 791 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Referral rates of intervention or conservative treatment in symptomatic severe AS (SAVR vs. TAVI vs. medical treatment) in different types of hospitals | 12 months
  The purpose of this study is to determine treatment pathways for patients with severe AS and to find out about the critical steps in this pathway with respect to the time-course and treatment decisions made.

SECONDARY OUTCOMES:
Transition of asymptomatic in symptomatic severe aortic stenosis (clinical evaluation of shortness of breath, chest pain and/or dizziness or syncope) | 12 months
  Time course for the transition from asymptomatic in symptomatic severe AS and analysis of multivariables predictors for the development of symptoms (based on echo data and comorbidities at baseline)
Outcomes (survival) (intervention vs. conservative treatment) | 12 months
  rates of death

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Balduss, Prof, Study Chair — University of Cologne; Norbert Frey, Prof, Study Chair — University of Kiel, Germany; Richard Steeds, Prof, Study Chair — Queen Elizabeth Hospital, Birmingham, UK; David Messika-Zeitoun, Prof, Study Chair — Bichat Hospital
Locations (2):
- Bichat Hospital Paris, Paris, France
- Department of Cardiology and Angiology, University of Kiel, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No
no sharing of individual patient data is planned

REFERENCES:
- [Derived] Rudolph TK, Messika-Zeitoun D, Frey N, Lutz M, Krapf L, Passefort S, Fryearson J, Simpson H, Mortensen K, Rehse S, Tiroke A, Dodos F, Mies F, Deutsch C, Kurucova J, Thoenes M, Bramlage P, Steeds RP; IMPULSE enhanced investigators. Severe aortic stenosis management in heart valve centres compared with primary/secondary care centres. Heart. 2023 May 26;109(12):944-950. doi: 10.1136/heartjnl-2022-321566. PMID 36657962
- [Derived] Rudolph TK, Messika-Zeitoun D, Frey N, Lutz M, Krapf L, Passefort S, Fryearson J, Simpson H, Mortensen K, Rehse S, Tiroke A, Dodos F, Mies F, Pohlmann C, Kurucova J, Thoenes M, Bramlage P, Steeds RP. Caseload management and outcome of patients with aortic stenosis in primary/secondary versus tertiary care settings-design of the IMPULSE enhanced registry. Open Heart. 2019 Jul 21;6(2):e001019. doi: 10.1136/openhrt-2019-001019. eCollection 2019. PMID 31413844